CLINICAL TRIAL: NCT04838756
Title: A Randomized, Single-blinded, Controlled Trial on the Efficacy of Mammography Screening With Artificial Intelligence - the MASAI Study
Brief Title: Mammography Screening With Artificial Intelligence (MASAI)
Acronym: MASAI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Unilabs (Unknown); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2020-04936
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Mammography Screening; Artificial Intelligence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants have the possibility to opt-out. If they do not opt-out, neither the participant nor the nurse performing the screen exam will know to what study arm the participant was allocated. The radiologist reading the screen exam will however not be blinded to allocation information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): AI-integrated mammography screening
  Interventions: Other: AI screening modality
- Control arm (Experimental): Conventional mammography screening (standard of care)
  Interventions: Other: Conventional screening modality

INTERVENTIONS:
Other: AI screening modality — Screen exam will be analysed with an AI system (Transpara, ScreenPoint, Nijmegen, The Netherlands) that assigns exams with a cancer-risk score from 1 to 10, as well as presenting CAD-marks at suspicious findings. Exams with risk score 1-9 will be single read and exam with score 10 will be double read. Risk scores and CAD-marks are provided to the reader(s). The reader(s) will decide whether to recall the woman for work-up or not (as per standard of care). In addition, exams with the highest 1% risk will by default be recalled with the exception of obvious false positives.
  Arms: Intervention arm
Other: Conventional screening modality — Screen exams will be read by two radiologists without the support of AI.
  Arms: Control arm

SUMMARY:
The purpose of this randomized controlled trial is to assess whether AI can improve the efficacy of mammography screening, by adapting single and double reading based on AI derived cancer-risk scores and to use AI as a decision support in the screen reading, compared with conventional mammography screening (double reading without AI).

DETAILED DESCRIPTION:
European guidelines recommend that mammography exams in breast cancer screening are read by two breast radiologists to ensure a high sensitivity. Double reading is, however, resource demanding and still results in missed cancers. Computer-aided detection based on AI has been shown to have similar accuracy as an average breast radiologist. AI can be used as decision support by highlighting suspicious findings in the image as well as a means to triage screen exams according to risk of malignancy.

Eligible women will be randomized (1:1) to the intervention (AI-integrated mammography screening) or control arm (conventional mammography screening). In the intervention arm, exams will be analysed with AI and triaged into two groups based on risk of malignancy. Low risk exams will be single read and high risk exams will be double read. The high risk group will contain appx. 10% of the screening population. Within the high-risk group, exams with the highest 1% risk will by default be recalled by the readers with the exception of obvious false positives. AI risk scores and Computer-Aided Detection (CAD)-marks of suspicious calcifications and masses are provided to the reader(s). In the control arm, screen exams are double read without AI (standard of care). Considering the interplay of number of interval cancers and workload, the study will be considered successful if the interval-cancer rate in the intervention arm is not more than 20% larger than in the control arm. If the interval-cancer rate is statistically and clinically significantly lower in the intervention arm than in the control arm, AI-integrated mammography screening will be considered superior to conventional mammography screening.

ELIGIBILITY:
Inclusion Criteria:

Women eligible for population-based mammography screening.

Exclusion Criteria:

None.

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
Interval-cancer rate | 43 months
  Women with interval cancer per 1000 screens

SECONDARY OUTCOMES:
Cancer-detection rate | 15 months
  Women with screen-detected cancer per 1000 screens
Recall rate | 15 months
  Number of recalls per 1000 screens
False-positive rate | 15 months
  Women with false positive per 1000 screens
Positive Predictive Value-1 | 15 months
  Women with cancer for all recalls
Sensitivity and specificity | 43 months
  True and false-positive rate
Cancer detection per cancer type | 19 months
  Screen detection of cancer in relation to cancer type, size and stage
Tumour biology of interval cancers | 43 months
  Characterization of interval cancers per type, size and stage
Screen-reading workload | 19 months
  Number of screen-readings and number of consensus meetings
Incremental cost-effectiveness ratio | 43 months
  The incremental cost-effectiveness ratio for AI-integrated mammography screening versus standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Lång, MD PhD, Principal Investigator — Region Skåne
Locations (1):
- Mammography Unit, Unilabs/Skane University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD could be considered to be shared in future collaborations.

REFERENCES:
- [Result] Lang K, Josefsson V, Larsson AM, Larsson S, Hogberg C, Sartor H, Hofvind S, Andersson I, Rosso A. Artificial intelligence-supported screen reading versus standard double reading in the Mammography Screening with Artificial Intelligence trial (MASAI): a clinical safety analysis of a randomised, controlled, non-inferiority, single-blinded, screening accuracy study. Lancet Oncol. 2023 Aug;24(8):936-944. doi: 10.1016/S1470-2045(23)00298-X. PMID 37541274
- [Result] Hernstrom V, Josefsson V, Sartor H, Schmidt D, Larsson AM, Hofvind S, Andersson I, Rosso A, Hagberg O, Lang K. Screening performance and characteristics of breast cancer detected in the Mammography Screening with Artificial Intelligence trial (MASAI): a randomised, controlled, parallel-group, non-inferiority, single-blinded, screening accuracy study. Lancet Digit Health. 2025 Mar;7(3):e175-e183. doi: 10.1016/S2589-7500(24)00267-X. Epub 2025 Feb 3. PMID 39904652
- [Derived] Gommers J, Hernstrom V, Josefsson V, Sartor H, Schmidt D, Hjelmgren A, Larsson AM, Hofvind S, Andersson I, Rosso A, Hagberg O, Lang K. Interval cancer, sensitivity, and specificity comparing AI-supported mammography screening with standard double reading without AI in the MASAI study: a randomised, controlled, non-inferiority, single-blinded, population-based, screening-accuracy trial. Lancet. 2026 Jan 31;407(10527):505-514. doi: 10.1016/S0140-6736(25)02464-X. PMID 41620232